CLINICAL TRIAL: NCT06466629
Title: The Optimal Timing of Vaccination in Pregnancy: a Multi-dimensional Mechanistic Approach to Measure Immune Responses in Pregnant Women
Brief Title: The Optimal Timing of Vaccination in Pregnancy
Acronym: MATIMMUNE
Status: Recruiting | Type: Observational
Sponsor: Elke Leuridan, MD, PhD (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Sponsor-Investigator, Elke Leuridan, MD, PhD, Principal Investigator, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Other Study IDs: cev005
Record Dates: First submitted 2022-11-16; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pertussis/Whooping Cough
MeSH Terms: conditions — Whooping Cough | interventions — adacel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Cord blood, breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Pregnant women vaccinated with Tdap vaccine between 16-18 weeks of gestation
  Interventions: Biological: Triaxis, Sanofi Pasteur
- Cohort 2: Pregnant women vaccinated with Tdap vaccine between 25-27 weeks of gestation
  Interventions: Biological: Triaxis, Sanofi Pasteur
- Cohort 3: Pregnant women vaccinated with Tdap vaccine between 34-36 weeks of gestation
  Interventions: Biological: Triaxis, Sanofi Pasteur

INTERVENTIONS:
Biological: Triaxis, Sanofi Pasteur — tetanus, diphtheria, acellular pertussis (aP) (Tdap) vaccine

SUMMARY:
The central aim of this study is to investigate the optimal timing of vaccination in pregnant women. Therefore, pregnant women will be vaccinated against pertussis at different timepoints and blood and breast milk samples will be taken at several timepoints. The main objectives are to assess the impact of timing on humoral and cellular immune responses in pregnant women, on antibody characteristics transferred across the placenta and on transplacental transport efficiency. The impact of maternal pertussis vaccination and timing of maternal pertussis vaccination on breastmilk antibody composition will also be investigated, as well as the impact of vaccination during pregnancy on the mucosal uptake of breastmilk IgA antibodies by the infant respiratory and gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* Willing to be vaccinated with a Tdap vaccine during pregnancy.
* Intend to be available for follow-up visits and phone call access until 6 months postpartum.
* Influenza and COVID-19 vaccination during pregnancy (as per Belgian recommendations) is allowed.

Exclusion Criteria:

* Vaccinated with an aP containing vaccine during the last 5 years
* Significant mental illness (e.g. schizophrenia, psychosis, major depression)
* Serious underlying immunological condition (e.g. immunosuppressive disease or therapy, human immunodeficiency virus (HIV) infection…).
* Systemic treatment with immune suppressive medication, including chronic steroid use of > 10 mg prednisone or equivalent.
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk.
* Previous severe reaction to any vaccine
* High risk for serious obstetrical complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female pregnant population within Flanders
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of antibody levels, subclass antibody levels, antibody glycosylation and antibody functionality in maternal blood after Tdap vaccination at different timings in pregnancy. | Before Tdap vaccination
Measurement of antibody levels, subclass antibody levels, antibody glycosylation and antibody functionality in maternal blood after Tdap vaccination at different timings in pregnancy. | One month after Tdap vaccination
Measurement of antibody levels, subclass antibody levels, antibody glycosylation and antibody functionality in maternal blood after Tdap vaccination at different timings in pregnancy. | At delivery
Measurement of antibody levels, subclass antibody levels, antibody glycosylation and antibody functionality in maternal blood after Tdap vaccination at different timings in pregnancy. | 6 months postpartum

SECONDARY OUTCOMES:
Measurement of cytokine levels and T-cell subsets in maternal blood after Tdap vaccination at different timings in pregnancy. | Before Tdap vaccination
Measurement of cytokine levels and T-cell subsets in maternal blood after Tdap vaccination at different timings in pregnancy. | One month after Tdap vaccination
Measurement of cytokine levels and T-cell subsets in maternal blood after Tdap vaccination at different timings in pregnancy. | At delivery
Measurement of cytokine levels and T-cell subsets in maternal blood after Tdap vaccination at different timings in pregnancy. | 6 months postpartum
Measurement of antibody levels in cord blood at delivery after Tdap vaccination at different timings in pregnancy to calculate the transport of antibodies across the placenta | At delivery
Measurement of antibody levels, subclass antibody levels, antibody glycosylation and antibody functionality in breastmilk after Tdap vaccination at different timings in pregnancy. | 6 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Vaccinopolis, Edegem, Antwerp, Belgium